CLINICAL TRIAL: NCT04730128
Title: Translation and Validation of the Hirschsprung and Anorectal Malformation Quality of Life (HAQL) Questionnaire in a Danish Hirschsprung Population
Brief Title: Translation and Validation of a Disease-specific Questionnaire for Hirschsprung's Disease in Danish Patients
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Kristina Gosvig, Principal Investigator, University of Southern Denmark
Other Study IDs: 011-2018-NQ
Record Dates: First submitted 2021-01-25; First posted 2021-01-29 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Hirschsprung Disease
Keywords: Hirschsprung Disease; Quality of Life; Translation and validation
MeSH Terms: conditions — Hirschsprung Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Hirschsprung and anorectal malformation quality of life (HAQL) questionnaire is a disease-specific quality of life questionnaire with 5 different elements (3 questionnaires for patients (categories: age 8-11, 12-16, and >17 years) and two questionnaires for parents of patients (categories: patients aged 8-11 and 12-16 years).

In the first part of this study, the questionnaires will be translated via forward-backward-translation, culturally adapted and evaluated for content validity.

In the second part of the study, the questionnaires will be validated in a cohort of all eligible Hirschsprung patients from Odense University Hospital from 1985-2014.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Hirschsprung's Disease between the years 1985-2014
* Age > 7 years
* Good Danish comprehension
* Signed informed consent

Exclusion Criteria:

* Inability to follow the procedures of the study, e.g. due to language problems, severe psychological disorders, dementia, etc.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Based on the ICD-10 code for Hirschsprung's disease, all patients with Hirschsprung's disease diagnosed in Odense University Hospital will be offered to participate in the study. The diagnosis must be registered between the years 1985-2014 and the patient must be > 7 years at the study initiation.
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Internal Consistency (IC) assessed by Cronbach's Alpha | Day 1

SECONDARY OUTCOMES:
Test-retest reliability assessed by intraclass-correlations coefficient | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense, Region Syddanmark, Denmark